CLINICAL TRIAL: NCT01257581
Title: Phase 2 Selection Trial of High Dosage Creatine and Two Dosages of Tamoxifen in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety and Efficacy Study of Creatine and Tamoxifen in Volunteers With Amyotrophic Lateral Sclerosis (ALS)
Acronym: SDALS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nazem Atassi (Other)
Collaborators: ALS Therapy Alliance (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor-Investigator, Nazem Atassi, Nazem Atassi, MD. MMSc., Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDALS-001
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's Disease; Amyotrophic Lateral Sclerosis; Creatine; Tamoxifen; Selection Design
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Creatine; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Creatine 30gm (Experimental): Creatine will be taken as a powder mixed into food or liquid twice a day. Volunteers in this arm will take a total of 30gm of creatine per day for 38 weeks. Volunteers will also take placebo capsules twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Creatine is a nutritional supplement and is not approved by the U.S. Food and Drug Administration (FDA) for treating ALS.
  Interventions: Drug: creatine
- Tamoxifen 40mg (Experimental): Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 40mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Tamoxifen is approved by the U.S. Food and Drug Administration (FDA) for breast cancer treatment but is not approved for treating ALS.
  Interventions: Drug: tamoxifen
- Tamoxifen 80mg (Experimental): Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 80mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Tamoxifen is approved by the U.S. Food and Drug Administration (FDA) for breast cancer treatment but is not approved for treating ALS.
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: creatine — creatine monohydrate powder
  Arms: Creatine 30gm
Drug: tamoxifen — Tamoxifen citrate capsules
  Other Names: Nolvadex, Istubal, Valodex
  Arms: Tamoxifen 40mg; Tamoxifen 80mg

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of high dose creatine and two dosages of tamoxifen treatment in amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare, neurodegenerative disorder that results in progressive wasting and paralysis of voluntary muscles. It is known that nerve cells called motor neurons die in the brains and spinal cords of people with amyotrophic lateral sclerosis (ALS). However, the cause of this cell death is unknown.

In this double blind, randomized, selection design trial, researchers will evaluate the safety and effectiveness of creatine and tamoxifen in volunteers with ALS. There are a large number of potential drugs that may improve the survival or slow down the disease progression in people with ALS. The current strategy is to test one drug at a time against placebo. "Selection Design" is a different type of study design. A Selection Design study uses multiple drugs to screen against each other and picks the winner to take to a larger study. This design can speed the search for effective drugs to treat ALS. In this Selection Design study, each volunteer will take one active study drug (creatine 30gm, tamoxifen 40mg, or tamoxifen 80mg) and one placebo.

Approximately 60 eligible volunteers with ALS will be recruited from multiple centers in the US that belong to the Northeast ALS Consortium (NEALS). Volunteers will be randomly assigned equally to the three treatment arms: creatine 30gm/day, tamoxifen 40mg/day and tamoxifen 80mg/day. Volunteers will take study treatment for 38 weeks. After screening and randomization, volunteers will be followed at weeks 4, 10, 18, 28 and week 38. A final telephone interview will occur at week 42 (off study drug).

ELIGIBILITY:
Inclusion Criteria:

* Familial or sporadic ALS.
* Disease duration from diagnosis no greater than 36 months at Screening Visit.
* Aged 18 years or older.
* Capable of providing informed consent and complying with trial procedures.
* Vital capacity (VC) equal to or more than 50% predicted normal value for gender, height and age at the Screening Visit.
* Not taking, or on a stable dose of riluzole (50mg bid) for at least 30 days prior to the Screening Visit.
* Women must not be able to become pregnant for the duration of the study (e.g., post menopausal for at least one year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and be non-lactating.

Exclusion Criteria:

* History of known sensitivity or intolerability to creatine monohydrate or tamoxifen citrate or to any other related compound.
* Prior exposure to creatine or tamoxifen within 30 days of the Screening Visit.
* Exposure to any investigational agent within 30 days of the Screening Visit.
* Use of coumarin anticoagulants (warfarin sodium), rifampin, aminoglutethimide, medroxyprogesterone, letrozole, or bromocriptine.
* Presence of any of the following clinical conditions: Clinical evidence of unstable medical or psychiatric illness at the Screening Visit; Screening aspartate aminotransferase (AST) > 3 times the upper limit of normal or serum creatinine > 1.5 mg/dl (133 umol/L); Permanent assisted ventilation or mechanical ventilation; or Lactating or have a positive serum pregnancy test at the Screening Visit.
* History of any of the following: blood clots including deep vein thrombosis, pulmonary embolism, and stroke, cataracts, renal problems, endometrial cancer, uterine sarcoma, or diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazem Atassi, MD, MMSc, Principal Investigator — Masaschusetts General Hospital, Boston, MA
Locations (9):
- United States (9):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Washington University at St. Louis, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Pennsylvania State University, Hershey Medical Center, Hershey, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Northeast ALS Consortium website — http://www.alsconsortium.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine 30gm: Creatine will be taken as a powder mixed into food or liquid twice a day. Volunteers in this arm will take a total of 30gm of creatine per day for 38 weeks. Volunteers will also take placebo capsules twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Creatine is a nutritional supplement and is not approved by the U.S. Food and Drug Administration (FDA) for treating ALS.
  creatine: creatine monohydrate powder
- Tamoxifen 40mg: Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 40mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Tamoxifen is approved by the U.S. Food and Drug Administration (FDA) for breast cancer treatment but is not approved for treating ALS.
  tamoxifen: Tamoxifen citrate capsules
- Tamoxifen 80mg: Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 80mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
  This is a blinded study, so neither participants nor study staff will know which treatment a volunteer is receiving.
  Tamoxifen is approved by the U.S. Food and Drug Administration (FDA) for breast cancer treatment but is not approved for treating ALS.
  tamoxifen: Tamoxifen citrate capsules
Period: Overall Study
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Started | 22 | 21 | 17
Completed | 17 | 18 | 11
Not Completed | 5 | 3 | 6
Not completed — Early Termination | 3 | 1 | 2
Not completed — Death | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Efficacy outcomes are adjusted for baseline differences in time from symptom onset to diagnosis, site of symptom onset, and VC.
Groups:
- Creatine 30gm: Creatine will be taken as a powder mixed into food or liquid twice a day. Volunteers in this arm will take a total of 30gm of creatine per day for 38 weeks. Volunteers will also take placebo capsules twice a day for 38 weeks.
- Tamoxifen 40mg: Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 40mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
- Tamoxifen 80mg: Tamoxifen will be taken as capsules twice a day. Volunteers in this arm will take a total of 80mg of tamoxifen per day for 38 weeks. Volunteers will also take placebo powder twice a day for 38 weeks.
- Total: Total of all reporting groups
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg | Total
Number analyzed (Participants) | 22 | 21 | 17 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.4) | 60.3 (10.6) | 56.3 (11.3) | 57.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 9 | 19
  Male | 16 | 17 | 8 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 21 | 17 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 20 | 17 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 17 | 60
Years from Symptom Onset to Screening [Mean (Standard Deviation); unit: years] | 2.8 (1.7) | 1.9 (1.4) | 2.0 (1.0) | 2.3 (1.5)
Years from Diagnosis to Screening [Mean (Standard Deviation); unit: years] | 1.3 (0.8) | 0.9 (0.8) | 1.0 (0.8) | 1.1 (0.8)
Years from Symptom Onset to Diagnosis [Mean (Standard Deviation); unit: years] | 1.6 (1.5) | 0.9 (0.8) | 1.0 (0.8) | 1.2 (1.1)
Baseline ALS Functional Rating Scale - Revised (ALSFRS-R) Total [Mean (Standard Deviation); unit: Score on a scale] — The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
  Score on a scale | 35.82 (7.20) | 36.19 (6.04) | 34.76 (6.56) | 35.65 (6.54)
Baseline VC% Predicted Max [Mean (Standard Deviation); unit: % of predicted max value] — The vital capacity (VC) (percent of predicted normal) was determined using the slow VC method. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percent of predicted normal.
  % of predicted max value | 90.64 (20.29) | 86.90 (13.92) | 81.71 (19.93) | 86.80 (18.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in ALS Functional Rating Scale - Revised (ALSFRS-R)
Description: Primary efficacy will be assessed by analyzing the mean rate of decline in the ALS Functional Rating Scale-Revised (ALSFRS-R) score over nine months. The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
scores on a scale | -0.905 [-1.292 to -0.518] | -0.983 [-1.336 to -0.630] | -0.743 [-1.259 to -0.227]

2. Secondary Outcome: Vital Capacity/Pulmonary Function Testing
Description: Secondary efficacy will be assessed by analyzing the change in the Slow Vital Capacity score over nine months. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percentage of predicted normal.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: Percentage of predicted max value
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
Percentage of predicted max value | -3.386 [-4.794 to -1.977] | -2.915 [-4.216 to -1.615] | -3.377 [-5.203 to -1.552]

3. Secondary Outcome: Tracheostomy-free Survival
Description: Secondary efficacy will be assessed by analyzing rate of tracheostomy-free survival at nine months.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
proportion of participants | 0.455 [0.276 to 0.679] | 0.286 [0.140 to 0.528] | 0.412 [0.222 to 0.675]

4. Secondary Outcome: Dose Adjustments
Description: These events were due to a double-blinded study design.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Number; unit: Number of Events due to Adverse Events
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
Number of Events due to Adverse Events
  Number of Creatine Reductions due to AEs | 6 | 3 | 0
  Tamoxifen Redutions due to AEs | 5 | 4 | 0
  Suspensions due to AEs | 9 | 1 | 2
  Discontinuations due to AEs | 10 | 5 | 4

5. Secondary Outcome: Lab Abnormal Reports by Treatment Assignment
Description: The safety data is summarized according to treatment arm. Total number of Adverse Events (AEs), AEs that cause study drug withdrawal and abnormal laboratory tests are compared among treatment arms. A lab abnormality was a result that was out of range and considered clinically significant by the site investigator.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Number; unit: Events
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
Events
  ALT (SGOT) | 0 | 1 | 0
  Creatinine | 4 | 0 | 0
  Glucose | 0 | 0 | 1
  Hematocrit | 1 | 0 | 0
  Lymphocytes | 1 | 0 | 0
  MCH | 1 | 0 | 0
  Neutrophils | 0 | 0 | 1
  Absolute Neutrophils | 0 | 0 | 1
  GFR Non-African American | 2 | 0 | 0
  Potassium | 0 | 0 | 1
  Red Blood Count (RBC) | 1 | 0 | 0
  White Blood Count (WBC) | 1 | 0 | 0

6. Secondary Outcome: Hand Held Dynamometry (HHD) Lower Z-score
Description: The HHD lower z-scores are means of z-scores for right and left knee extension, knee flexion, hip flexion, and ankle dorsiflexion with z-scores calculated relative to the baseline mean and standard deviation strength of each muscle group across all participants.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
Z-score | -0.094 [-0.127 to -0.061] | -0.067 [-0.096 to -0.039] | -0.016 [-0.052 to 0.020]

7. Secondary Outcome: HHD Lower % Baseline
Description: HHD % baseline measures are mean percent change for right and left knee extension, knee flexion, hip flexion, and ankle dorsiflexion from each participant's baseline.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
percent change | -9.258 [-13.118 to -5.399] | -6.711 [-10.302 to -3.121] | -2.897 [-7.440 to 1.646]

8. Secondary Outcome: HHD Upper Z-score
Description: The HHD upper z-scores are means of z-scores for right and left shoulder flexion, elbow extension, elbow flexion, write extension and first dorsal interosseous muscles with z-scores calculated relative to the baseline mean and standard deviation strength of each muscle group across all participants.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
Z-score | -0.103 [-0.159 to -0.048] | -0.089 [-0.142 to -0.037] | -0.039 [-0.105 to 0.027]

9. Secondary Outcome: HHD Upper % Baseline
Description: The HHD % baseline measures are mean percent change for shoulder flexion, elbow extension, elbow flexion, wrist extension, and first dorsal interosseous muscles from each participant's baseline.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
percent change | -8.451 [-11.726 to -5.175] | -7.720 [-10.697 to -4.743] | -4.515 [-8.063 to -0.968]

10. Secondary Outcome: Accurate Test of Limb Isometric Strength (ATLIS) Lower Percentage of Predicted Normal (PPN)
Description: The ATLIS PPN measures are percentages of predicted normal strength based on age, gender, height, and weight using normative data.
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: percentages of predicted normal strength
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
percentages of predicted normal strength | -2.098 [-3.931 to -0.266] | -2.375 [-4.441 to -0.310] | -0.491 [-2.759 to 1.776]

11. Secondary Outcome: ATLIS Upper Percentage of Predicted Normal (PPN)
Description: as for outcome 10
Time Frame: 38 weeks of treatment followed by a telephone interview at 42 weeks.
Measure: Mean (95% Confidence Interval); unit: percentages of predicted normal strength
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Number analyzed (Participants) | 22 | 21 | 17
percentages of predicted normal strength | -1.932 [-4.112 to 0.249] | -1.845 [-4.084 to 0.393] | 0.436 [-2.143 to 3.016]

ADVERSE EVENTS:
Arm/Group | Creatine 30gm | Tamoxifen 40mg | Tamoxifen 80mg
Serious Adverse Events (participants affected / at risk) | 6/22 | 3/21 | 5/17
Other Adverse Events (participants affected / at risk) | 21/22 | 17/21 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine 30gm (N=22) | Tamoxifen 40mg (N=21) | Tamoxifen 80mg (N=17)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine 30gm (N=22) | Tamoxifen 40mg (N=21) | Tamoxifen 80mg (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7) | 5 (5) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (8) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 4 (4) | 2 (3)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Application Site Rash (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (2) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 4 (4) | 7 (7)
Oedema Peripheral (General disorders) | 4 (5) | 2 (2) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 3 (3)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vital Capacity Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5) | 2 (4) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (7) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Contractions Involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peroneal Nerve Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Affect Lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 4 (4)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mole Excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes